CLINICAL TRIAL: NCT06920212
Title: Clinical Safety and Efficacy of FMT in the Treatment of Alzheimer's Disease
Brief Title: Clinical Safety and Efficacy of Fecal Microbiota Transplantation (FMT) in the Treatment of Alzheimer's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Dean of the hospital, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-AD
Record Dates: First submitted 2025-03-31; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMT (Experimental)
  Interventions: Procedure: FMT capsule

INTERVENTIONS:
Procedure: FMT capsule — Fecal microbiota transplantation (FMT) is a method for treating imbalances in the intestinal microbiota. Its basic principle involves extracting a portion of feces from a healthy individual that contains a diverse population of beneficial bacteria, processing it, and transplanting it into the digestive system of the recipient to restore a balanced intestinal microbiota.

SUMMARY:
To investigate the clinical safety and efficacy of FMT in AD patients, as well as the changes in the gut microbiota of AD patients before and after FMT.

ELIGIBILITY:
Inclusion Criteria:

* The patients (aged 50-85 years) exhibited cognitive decline persisting for over six months;
* Primarily characterized by recent memory impairment and accompanied by reduced daily living abilities;
* MMSE scores ranging from 3 to 26;
* MRI findings revealed atrophy in the medial temporal lobe, hippocampus, and cerebral cortex, along with widened sulci and fissures.

Exclusion Criteria:

* Patients were excluded if they had severe visual, hearing, or language impairments;
* Tumors;
* hepatic/renal dysfunction.
* with conditions mimicking AD symptoms-such as normal pressure hydrocephalus, vascular dementia (VD or VaD);
* Parkinson's disease dementia (PDD)-were also excluded;
* patients who had participated in clinical drug trials within the past 30 days or consumed folate and vitamin B12 at doses exceeding twice the recommended intake were ineligible.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoints | 0, 1month, 2months, 3months, 6months
  Changes in scores on the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)
Efficacy endpoints | 0, 1month, 2months, 3months, 6months
  Changes in scores on Mini-Mental State Examination (MMSE).
Efficacy endpoints | 0, 1month, 2months, 3months, 6months
  Changes in scores on Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADAS-CGIC).
Efficacy endpoints | 0, 1month, 2months, 3months, 6months
  Changes in scores on Alzheimer's Disease Activities of Daily Living Scale (ADAS-ADL)
Changes in gut microbiota | 0, 1month, 2months, 3month, 6months
  Gut metagenomic sequencing was performed to conduct OTU (Operational Taxonomic Unit) clustering and taxonomic analysis, comparing alterations in patients' intestinal flora before and after FMT.

CONTACTS AND LOCATIONS:
Locations (1):
- Le Wang, Shanghai, China